CLINICAL TRIAL: NCT04280614
Title: Day Hospital Treatment of Emotional Dysregulation: A Quantitative Analysis
Brief Title: Day Hospital Treatment of Emotional Dysregulation
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Daryl Croft, Principal Investigator, University of Manitoba
Other Study IDs: H2019:485
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Emotional Dysfunction
MeSH Terms: interventions — Dialectical Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Dialectical behaviour therapy (DBT) — DBT is based on the behavioural therapy principals focusing on four main modules: mindfulness, interpersonal effectiveness, emotional regulation and distress tolerance. The therapy is taught in a group and individual therapy model with coaching during periods of crisis. CBT is a standard model of therapy similar to DBT but is more direct in focusing clients on changing maladaptive behaviours or thoughts to effectively manage difficult emtions.
  Other Names: cognitive behaviour therapy (CBT)

SUMMARY:
Objective: The goal of this proposed research project is a quantitative analysis of a day hospital program designed to treat persons with emotional dysregulation.

Background: The Short-term Assessment and Treatment (STAT) program has been operating at Health Sciences Center, Winnipeg, Manitoba for many decades. The STAT program is based on the principles of dialectical and cognitive behavior therapy. The STAT program is a five week day hospital program employing multi-modal treatment methods to treat patients with emotional dysregulation. The literature provides evidence of numerous treatment models with varying effectiveness for this population of patients. The STAT program hasn't had a quantitative analysis of its treatment model.

Problem Statement: Is the 5 week day hospital treatment model developed and employed by the STAT program effective in improving the mental health of participants admitted to the program?

DETAILED DESCRIPTION:
Research on brief therapeutic interventions for those diagnosed with BPD have often involved a year or more of treatment in an outpatient, inpatient or partial hospitalization setting. The goal of this research proposal is to examine if a 5-week day hospital treatment program at a tertiary hospital within Shared Health can demonstrate effective amelioration of subject symptoms on a number of measures.

As noted in the introduction there is significant public health considerations associated with persons living with borderline personality disorder pathology. Evidence-based public health should be informed by practice-based evidence stemming from the rigorous evaluation of relevant natural experiments. Due to logistic and ethical considerations a randomized control trial isn't feasible. Given these considerations, the proposed research design is a naturalistic pre- post-intervention with no control group. Although causality cannot be determined in a naturalistic design, methodological rigour employed will mitigate the impact of outside variable from invalidating the results obtained from the proposed research. Participants data will be collected at two times and the data from the same individual will be compared focusing on differences between pre- and post-intervention. The benefit in the longitudinal design is the potential to control for temporal or secular changes observed in the outcome. A challenge in interpreting randomized control trials is potential biases that impact external validity and reduce the ability of the researchers to generalize the outcomes associated with an intervention. Naturalistic studies can reduce the impact of confounding variable by identifying and controlling potential variables, such as socio-economic factors.

Sample Characteristics and Selection Participants are referred to the STAT program through emergency room consultations, family physician referrals and from psychiatrists working in the community, outpatient department or during an inpatient admission. Participants are individuals 18 years and older.

Although participants in the STAT program are primarily females there is no exclusion criteria based on gender. These participants are assigned a therapist who will complete a psychiatric interview and review a self-report each participant is required to complete prior to the initial interview. Potential participants will meet with a psychiatrist to review the information gathered in the therapist interview and determine if the client will be admitted to the STAT day hospital program. Participants are accepted if they meet admission criteria as determined by the psychiatrist. Participants are excluded if they have a diagnosis of antisocial personality disorder, criminal charges, or significant substance abuse. Participants are required to formulate behaviour-oriented goals to work on while participating in the STAT program. Participants are not admitted to the program if they do not formulate treatment goals. Potential participants referred from one of the above noted sources are assigned to a therapist each Tuesday at a weekly meeting of the STAT program staff. The therapist will contact the individual and arrange a date for an initial interview. If a therapist is unable to reach an individual by phone, a letter with the date for an appointment is mailed along with the self-report questionnaire each client is expected to complete for the first interview with the therapist. The self-report materials include a series of questions to elicit a social history of the individual along with current stressors and self-identified problems. The assessment process involves roughly two appointments with the therapist and an additional appointment with the psychiatrist requiring roughly three weeks to complete. Participants will be given a letter of invitation outlining the research project as well as the SCL-90-R and DERS psychometric questionnaires. Individuals will be asked to complete the SCL-90-R and DERS at the beginning of their first appointment if they agree to participate in the research project.

Once an individual is accepted to the STAT Program, they are placed on the waiting list for a period of roughly four to six weeks. During that period, the therapist will meet with clients roughly two times to assist in formulating treatment goals and develop a therapeutic rapport. While a client is admitted to the program and participating in the groups, they are also seen by their assigned therapists on a weekly basis for an individual therapy session. Individual sessions with the therapist assist participants in understanding the psychoeducation group learning materials, assist with homework, and to process current stressors.

The participants will complete the Symptom Checklist-90-Revised (SCL-90-R) and Difficulties in Emotion Regulation Scale (DERS) prior to the first interview. Participants will be re-administered the SCL-90-R and DERS following completion of the 5-week treatment.

Program Description The Short-term Assessment and Treatment (STAT) program is a day hospital program operated at Health Sciences Center in Winnipeg, Manitoba. The STAT program operates a 5 week continuously running treatment program. Clients are admitted to and complete the program weekly. Similarly, other researchers have had participant entering the program at different points in the skill training and found no interaction effect and didn't significantly influence the participants' frequency or type of skills practised. The number of clients in the group is roughly 15 - 18. The STAT program employs a multidisciplinary team comprised of social workers, an occupational therapist, several nurses and psychiatrists.

The STAT program is comprised of psychoeducation and psychotherapy groups, and individual therapy with an assigned therapist. Clients attend morning and afternoon groups daily for the 5-week duration of the program. Groups are scheduled for 1 hr 30 min with an hour break for lunch. Two therapists lead each group and rotate through groups on a predetermined schedule. Psychoeducation groups are informed by the principles of DBT and CBT. Many of the skills taught are directly taken from Dr. M. Linehan's DBT skills training manual. Psychoeducation is taught in the morning with the assigned module handed out at the beginning of the week. There are six psychoeducation topics that clients will be taught during the course of treatment. One of five topics is introduced on Monday and mindfulness is taught each Friday. These topics are: Distorted Thinking, Anger Being Effective, Communication and Assertiveness, Goal-Setting and Self-Esteem. A new skill related to the mindfulness psychoeducation module is introduced each Friday. Participants are given daily reading material and homework to complete related to the weekly topic. Participants are asked to share daily from their homework in the group.

Many people with emotional struggles cope by engaging in self-injurious behaviours. Monday afternoon group focuses on the principles of Harm Reduction. Harm reduction groups teach the principles of stages of change, effective coping, and distress tolerance skills taught in DBT. Psychotherapy groups occur in the afternoon between Tuesday and Thursday. Participants are required to "check-in" at the beginning of group with a topic they would like to discuss.

Procedure As outlined above, participants will be given a letter of invitation outlining the research project a demographics questionnaire, the SCL-90-R and the DERS psychometric questionnaires. Individuals will be asked to complete the SCL-90-R and DERS at their first appointment if they agree to participate in the research project. The two questionnaires will be handed into the therapist along with the original copy of their signed Informed Consent. Participants will retain a copy of the informed consent letter along with the letter of invitation. The therapists will have adhesive identifiers to correspond the pre- and post-intervention self-report questionnaire to the participant. The therapist will affix an identifier to the envelope indicating the anonymous participant envelop contains preintervention self-report data. The therapist will code if the patient participated in psychoeducation and psychotherapy groups or just the psychoeducation groups. The rationale for the distinction is to control the confounding variable of differences in the treatment a participant will receive. For the purposes of this research project only participants that attend both psychoeducation and psychotherapy groups will be examined. Attrition will be accounted for and those participants will be compared with treatment completers to examine potential significant differences between these groups. Attrition will be identified by only having a pre-intervention self-report surveys completed. The participant will be given a card with the identifier number and the therapist will affix the third adhesive identifier to an envelope for the post-intervention assessment. Participants will be re-administered the SCL-90-R and DERS following completion of the 5-week treatment. The participants will be given the two instruments on the last day in the program to complete. The therapist will ask the participants if they have the card given to them with identifier affixed when they completed the pre-intervention questionnaire. The participants will be given the corresponding post-intervention envelope containing the SCL-90-R and DERS surveys. The participants will hand in the completed questionnaires to their therapist. The goal will be to solicit 60 clients to the research project.

Anticipated Outcomes The author expects that there will be an improvement in global severity index, improvement of emotion regulation, and a reduction hostility and improved interpersonal relationships as self-reported. Literature has reported attrition rates upwards of 30% for treatment programs with those who have borderline personality disorder attributed to a lack of motivation, interpersonal conflict, difficulties with emotional distress, substance use, suicide attempts and antisocial personality disorder. The STAT program model may reduce the attrition rate because potential participants with significant substance abuse and an antisocial personality disorder are excluded from participating in the program. Researchers have noted attrition was related to treatment characteristics and life circumstances. The STAT program will not admit participants that don't have housing, stable finances such as employment insurance, and a family physician. Many treatments including standard DBT and mentalization-based therapy are also lengthier potentially making commitment for participants more difficult. Related to the admission criteria and the brief structure of STAT program the author expects the rate of attrition to be below the 30% rate noted above.

Proposed Data Analysis

A repeated measures t-test or an ANOVA data analysis will be used to determine if there is a predicted significant improvement in participants self-reports between pre- and post-intervention. An exploratory correlation data analysis will be used to examine if there are differences between participants that complete the STAT program versus those that don't complete the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older

Exclusion Criteria:

* declined by the STAT Program

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are referred to the STAT program through emergency room consultations, family physician referrals and from psychiatrists working in the community, outpatient department or during an inpatient admission. Most potential participants live within the catchment of Winnipeg.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Self-harm, emotional distress, depression, anxiety | Roughly 8 weeks.
  The Symptom-Checklist-90-Revised is a psychometric measure used in research and clinical settings in measurement of outcomes related to treatment. It measures global severity of mental illness, positive symptom distress index, positive symptom total as well as nine dimensions of psychopathology on a 0 - 4 scale. Previous research studies on therapeutic interventions involving BPD participants have used the SCL-90-R to measure outcome. The SCL-90-R will be used to assess if the participants self-report a decrease in the severity of global indices of mental illness and nine specific psychopathology factors. Gratz and Roemer (2004) developed the Difficulties in Emotion Regulation Scale (DERS), a 36 item self-report survey to assess emotion dysregulation on six domains. DERS has good test-retest reliability and high internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It's unclear to what extent my thesis will be shared. The intent at this juncture is to present the data as a whole and not identify individual participant data in dissemination. Further discussion with my thesis advisor and the thesis advisory team is ongoing.